CLINICAL TRIAL: NCT05223491
Title: En Bloc Transurethral Resection of Non-muscle Invasive Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jørgen Bjerggaard Jensen (Other)
Collaborators: University of Aarhus (Other); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, Professor, DMSc, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: En Bloc
Record Dates: First submitted 2022-01-07; First posted 2022-02-04 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2024-09

CONDITIONS: Non-muscle Invasive Bladder Cancer
Keywords: en bloc; TURB
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- En Bloc (Experimental): The bladder tumour will be resected en bloc and removed in total, if possible.
  Interventions: Procedure: En Bloc resection
- Conventional TURB (Active Comparator): The bladder tumour will be removed by conventional piecemeal resection.
  Interventions: Procedure: Conventional TURB

INTERVENTIONS:
Procedure: En Bloc resection — Tumour is resected and removed from the bladder in one piece, if possible.
  Arms: En Bloc
Procedure: Conventional TURB — Tumour is resected piecemeal.
  Arms: Conventional TURB

SUMMARY:
Aim: To compare the surgical method of En Bloc resection to the conventional transurethral resection of non-muscle invasive bladder cancer (NMIBC) in terms of complete removal of tumour, specimen quality, and pathological certainty.

Background: NMIBC is a common disease with a 5-year recurrence rate reported as high as 64%. The cornerstone in the treatment of NMIBC is transurethral resection (TURB) where the tumour is dissected in pieces, removed from the bladder, and pathologically examined for potential muscle invasion. As the tumour is fragmented before removal, the method violates basic oncological principles and compromises pathological examination. Hence, TURB is possibly part of the mechanism causing recurrences. En Bloc resection (EBR), where the tumour is removed in toto, can potentially overcome the flaws of conventional TURB, but large randomized trials are needed.

Methods: This project will be a multicentre randomised controlled clinical trial comparing EBR to conventional TURB. Patients with suspected NMIBC tumours with largest tumour diameter ≥1cm and ≤6cm will be randomised to either the intervention group, thus undergoing EBR, or the control group, undergoing conventional TURB. The investigators intend to include 220 patients in total, 110 patients in each group. The RCT will be initiated in 2022.

Perspectives: If EBR can be shown to remove bladder tumours with better pathological quality and certainty, this could potentially spare patients from undergoing surgeries in the future, thereby reducing costs for both patients and society.

ELIGIBILITY:
Inclusion Criteria:

* Demographics: all BMI, smokers and non-smokers
* Primary, papillary, non-solid bladder tumour visualised by flexible cystoscopy
* Tumour diameter measured on CT-scan ≥2cm ≤6cm at largest diameter
* Ability to fully comprehend the information provided and comply with protocol
* Signed consent form
* Patients with multiple tumours can be included if it seems feasible to resect them in one procedure

Exclusion Criteria:

* Clinically suspected muscle invasive bladder cancer (invasion in to bladder muscle or extravesical extension visible on CT or solid tumour without papillary elements seen at cystoscopy)
* Tumour located in a bladder diverticulum
* Investigating physician concludes that en bloc resection is not technically possible
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Unaltered pathological T-stage | 4 months
  Proportion of patients with unaltered pathological T-stage following central pathology revision, reTURB, or cystectomy compared to initial T-stage description from TURB.

SECONDARY OUTCOMES:
Detrusor muscle in specimen | Within one week from surgery
  Prevalence of detrusor muscle in specimen by pathological examination
Recurrence free survival | 4 months
  Proportion of patients with recurrences at 4 months follow-up cystoscopy

CONTACTS AND LOCATIONS:
Locations (11):
- Denmark (7):
  - Department of Urology, Aalborg University Hospital, Aalborg
  - Department of Urology, Aarhus University Hospital, Aarhus
  - Department of Urology, Herlev Hospital, Herlev
  - Department of Urology, Regional Hospital Gødstrup, Holstebro
  - Department of Urology, Odense University Hospital, Odense
  - Department of Urology, Zealand University Hospital, Roskilde
  - Dept. of Urology, Hospital Lilelbælt, Vejle, Vejle
- Dept. of Urology, North Estonia Medical Centre, Tallinn, Estonia
- Dept. of Urology, Turku University Hospital, Turku, Finland
- Urological Center, Paula Stradina Clinical University Hospital, Riga, Latvia
- Department of Urology, Vestfold Hospital, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: No